CLINICAL TRIAL: NCT05075408
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of Nemolizumab in Subjects With Chronic Kidney Disease With Associated Moderate to Severe Pruritus
Brief Title: To Evaluate the Efficacy and Safety of Nemolizumab for 12 Weeks in Participants With Chronic Kidney Disease With Associated Moderate to Severe Pruritus
Acronym: NIKAIA 1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.06.SPR.204358; 2021-004766-35 (EudraCT Number)
Record Dates: First submitted 2021-09-30; First posted 2021-10-12 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease Associated Moderate to Severe Pruritus
Keywords: Chronic Kidney Disease; Moderate to Severe Pruritus; Nemolizumab; CD14152
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — nemolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: This was a double-blind study. The randomization code remained blinded to all participants, study sites personnel and Sponsor/CRO study team members until completion of the study and after the study database had been locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nemolizumab 30 mg (Experimental)
  Interventions: Drug: Nemolizumab
- Nemolizumab 60 mg (Experimental)
  Interventions: Drug: Nemolizumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nemolizumab — Participants received a loading dose of 60 mg nemolizumab at Baseline followed by 2 Subcutaneous (SC) injections for a total dose of 30 mg nemolizumab once every 4 weeks i.e. at Week 4 and Week 8.
  Other Names: CD14152
  Arms: Nemolizumab 30 mg
Drug: Nemolizumab — Participants received 2 SC injections of 30 mg nemolizumab once every 4 weeks i.e. at Week 4 and Week 8.
  Other Names: CD14152
  Arms: Nemolizumab 60 mg
Drug: Placebo — Participants received 2 SC injections of 30 mg placebo-matched to nemolizumab once every 4 weeks i.e. at Week 4 and Week 8.
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy of nemolizumab compared to placebo at reducing the intensity of pruritus after a 12-week treatment period in adult hemodialysis participants with moderate to severe pruritus.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged >= 18 years at the screening visit.
2. Had end-stage kidney disease (ESKD) and had been on hemodialysis three times per week for at least three months prior to the start of screening.

   Note 1: Participants who required an occasional additional hemodialysis treatment to manage fluid overload might be enrolled as long as it was anticipated that no more than one such treatment would be required in any given week.

   Note 2: Participants had received in-home hemodialysis might participated as long as they had switched to in-center hemodialysis at least two weeks prior to screening and plan to remain on in-center hemodialysis for the duration of the study.
3. Hemodialysis participants meeting the Kidney Outcome Quality Initiative Guidelines of hemodialysis adequacy within 60 days of screening, two:

   •Single-poolsKt/V measurements of at least 1.2.
4. Pruritus for >= three months (documented pruritus with no etiology identified other than CKD by medical record, previous physician's letter/statement, or a written conversation of site investigators based on the medical history obtained from the participant).
5. WI NRS score >= 5.0 at the screening and baseline visit. Screening WI NRS score would be determined by a single WI NRS assessment (score ranging from 0 to 10) for the 24-hour period immediately preceding the screening visit. Baseline WI NRS score would be determined based on the weekly average of daily WI NRS scores (score ranging from 0 to 10) during the seven days immediately preceding baseline (rounding was not permitted). A minimum of four daily scores out of the seven days immediately preceding baseline was required for this calculation.
6. Women of childbearing potential (WOCBP) (i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile) must agreed either to commit to true abstinence throughout the study and for 12 weeks after the last study drug injection, when this was in line with the preferred and usual lifestyle of the participant, or to use an adequate and approved method of contraception throughout the study and for 12 weeks after the last study injection.

   Adequate and approved methods of contraception applicable for the participant and/or her partner were defined below:
   * Progestogen-only oral hormonal contraception.
   * Combination of male condom with cap, diaphragm, or sponge with spermicide (double-barrier methods).
   * Combined (estrogen- and progestogen-containing) oral, intravaginal, or transdermal hormonal contraception.
   * Injectable or implanted hormonal contraception.
   * Intrauterine devices or intrauterine hormone releasing system.
   * Bilateral tubal ligation or tube insert (such as the Essure system) at least three months before the study.
   * Bilateral vasectomy of partner at least three months before the study.
7. Women were considered to be of non-childbearing potential if they meet one of the following criteria:

   * Absence of menstrual bleeding for one year prior to screening without any other medical reason, confirmed with follicle stimulating hormone (FSH) level in the postmenopausal range.
   * Documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy at least three months before screening.

   Note: Bilateral tubal ligation was not accepted as reason for non-childbearing potential.
8. Participant was willing and able to comply with all time commitments and procedural requirements of the clinical study protocol.
9. Understands and signs an informed consent form (ICF) before any investigational procedure(s) were performed.

Exclusion Criteria:

1. Body weight less than (<) 30 kg.
2. Pruritus caused by a concomitant condition unrelated to ESKD (e.g., dermatologic or systemic disorders such as, but not limited to atopic dermatitis (AD), psoriasis, prurigo nodularis (PN), Chronic T- cell Lymphoma, Leukemia or cholestatic liver disease).
3. Localized itch of only the palms of the hands and/or soles of the feet.
4. Pruritus present only during hemodialysis session.
5. History of or anticipated non-compliance with hemodialysis (i.e, such that it would adversely affect the conduct of the study or significantly change dialysis adequacy during the study) in the opinion of the investigator.
6. New York Heart Association Class IV symptoms or myocardial infarction within three months prior to screening.
7. History of stroke or transient ischemic attack within six months prior to screening.
8. Participants meeting one or more of the following criteria at screening or baseline:

   * Had an exacerbation of asthma requiring hospitalization in the preceding 12 months.
   * Reporting asthma that had not been well-controlled (i.e. symptoms occurring on greater than (>) two days per week, night time awakenings two or more times per week, or some interference with normal activities) during the preceding three months.
   * Asthma Control Test (ACT) <= 19 (only for participants with a history of asthma).
9. Cutaneous infection within one week before the baseline visit, any infection requiring treatment with oral or parenteral antibiotics, antivirals, antiparasitics or antifungals within two weeks before the baseline visit.
10. Any confirmed or suspected coronavirus disease (COVID-19) infection within two weeks before the screening or baseline visit. Participants might be rescreened after the infection had resolved. Resolution of COVID-19 infection could be confirmed by recovery assessment methods, as described in the protocol.
11. Positive serology results (hepatitis B surface antigen [HbsAg] or hepatitis B core antibody [HbcAb], hepatitis C [HCV] antibody with positive confirmatory test for hepatitis C virus [HCV] (e.g., HCV polymerase chain reaction [PRC]), or human immunodeficiency virus [HIV] antibody) at the screening visit.

    Note: Participants with a positive HbcAb and a negative HbsAg could be included in this clinical study if hepatitis B surface antibody was positive (considered immune after a natural infection or vaccination). Participants who were positive for HCV antibody and negative for HCV RNA might be enrolled.

    In the event of rescreening, the serology tests results (e.g., HBV, HCV, HIV) from the previous screening could be used by the investigator to assess the eligibility of rescreened participants if those tests were performed within six weeks prior to the baseline visit.
12. Known active or untreated latent tuberculosis (TB) infection or history of either untreated or inadequately treated active or latent TB according to the local applicable guidelines.

    Note: Participants who had a documented history of completion of an appropriate TB treatment regimen for latent or active TB with no history of re-exposure to TB since their treatment was completed were eligible to participate in the study.
13. Known or suspected immunosuppression beyond that expected due to end-stage kidney disease and its comorbidities or unusually frequent, recurrent, severe, or prolonged infections as per investigator judgment.
14. History of lymphoproliferative disease or history of malignancy of any organ system within the last five years, except for (1) basal cell carcinoma, squamous cell carcinoma in situ (Bowen's disease), or carcinomas in situ of the cervix that had been treated and had no evidence of recurrence in the last 12 weeks before the baseline visit, or (2) actinic keratoses that had been treated.
15. Pregnant women (positive serum pregnancy test result at any visits), breastfeeding women, or women planning a pregnancy during the clinical study.
16. In the opinion of the investigator the participant had any medical or psychological condition that could pose undue risk to the participant, prevent study completion, or adversely affect the validity or interpretability of the study measurements or interfered with study assessments.
17. Any clinically relevant laboratory abnormalities, such as but not limited to elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) (>3 * upper limit of normal [ULN]) in combination with elevated bilirubin (>2 * ULN), during the screening period that might put the participant at significant risk according to the investigator's judgment, if he/she participated in the clinical study.
18. Planned or expected major surgical procedure during the clinical study, including a scheduled kidney transplant during the study.
19. Had not adhered to the restrictions in the selected medications prior to screening or was not expected to be compliant with restrictions during the study.
20. Requiring rescue therapy for pruritus during the screening period or expected to require rescue therapy within 4 weeks following the Baseline visit.
21. Previous treatment with nemolizumab.
22. History of hypersensitivity (including anaphylaxis) to an immunoglobulin product (plasma-derived or recombinant, e.g. monoclonal antibody) or to any of the study drug excipients.
23. Currently participating or participated in any other study of an investigational drug or device, within the past four weeks (or five half-lives of the investigational medication, whichever was longer) before the screening visit.
24. History of alcohol or substance abuse within six months of the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (64):
- United States (47):
  - Galderma Investigational Site 9989, Bakersfield, California
  - Galderma Investigational Site 9991, Glendale, California
  - Galderma Investigational Site 7018, Glendale, California
  - Galderma Investigational Site 7015, La Palma, California
  - Galderma Investigational Site 9996, Los Angeles, California
  - Galderma Investigational Site 9978, Lynwood, California
  - Galderma Investigational Site 7017, Riverside, California
  - Galderma Investigational Site 9973, Tarzana, California
  - Galderma Investigational Site 7028, Victorville, California
  - Galderma Investigational Site 9964, Victorville, California
  - Galderma Investigational Site 7003, Whittier, California
  - Galderma Investigational Site 9971, Denver, Colorado
  - Galderma Investigational Site 9988, Bloomfield, Connecticut
  - Galderma Investigational Site 9980, Middlebury, Connecticut
  - Galderma Investigational Site 9970, Boca Raton, Florida
  - Galderma Investigational Site 7037, Coral Gables, Florida
  - Galderma Investigational Site 7026, Hollywood, Florida
  - Galderma Investigational Site 9965, Miami, Florida
  - Galderma Investigational Site7016, Miami, Florida
  - Galderma Investigational Site 7032, Sanford, Florida
  - Galderma Investigational Site 7004, Tampa, Florida
  - Galderma Investigational Site 7025, Tampa, Florida
  - Galderma Investigational Site 7027, Columbus, Georgia
  - Galderma Investigational Site 9983, Overland Park, Kansas
  - Galderma Investigational Site 9972, Wichita, Kansas
  - Galderma Investigational Site 9963, Roseville, Michigan
  - Galderma Investigational Site 7020, Edina, Minnesota
  - Galderma Investigational Site 9982, Minneapolis, Minnesota
  - Galderma Investigational Site 7035, Kansas City, Missouri
  - Galderma Investigational Site 9962, Las Vegas, Nevada
  - Galderma Investigational Site 7038, Fresh Meadows, New York
  - Galderma Investigational Site 9998, Great Neck, New York
  - Galderma Investigational Site 9995, The Bronx, New York
  - Galderma Investigational Site 7007, Winston-Salem, North Carolina
  - Galderma Investigational Site 9992, Roseburg, Oregon
  - Galderma Investigational Site 9999, Spartanburg, South Carolina
  - Galderma Investigational Site 9967, Chattanooga, Tennessee
  - Galderma Investigational Site 7039, Arlington, Texas
  - Galderma Investigational Site 7040, Dallas, Texas
  - Galderma Investigational Site 9966, El Paso, Texas
  - Galderma Investigational Site 9977, Greenville, Texas
  - Galderma Investigational Site 7011, Houston, Texas
  - Galderma Investigational Site 7022, McKinney, Texas
  - Galderma Investigational Site 7010, San Antonio, Texas
  - Galderma Investigational Site 7019, The Woodlands, Texas
  - Galderma Investigational Site 9968, Norfolk, Virginia
  - Galderma Investigational Site 9969, Wauwatosa, Wisconsin
- Hungary (5):
  - Galderma Investigational Site 6301, Budapest
  - Galderma Investigational Site 6304, Kecskemét
  - Galderma Investigational Site 6305, Miskolc
  - Galderma Investigational Site 6310, Szentes
  - Galderma Investigational Site 6298, Szombathely
- Poland (4):
  - Galderma Investigational Site 6294, Brodnica
  - Galderma Investigational Site 6296, Lodz
  - Galderma Investigational Site 6293, Olkusz
  - Galderma Investigational Site 6297, Wroclaw
- Spain (8):
  - Galderma Investigational Site 6309, Alcobendas
  - Galderma Investigational Site 6292, Córdoba
  - Galderma Investigational Site 5580, L'Hospitalet de Llobregat
  - Galderma Investigational Site 5171, Madrid
  - Galderma Investigational Site 6190, Madrid
  - Galderma Investigational Site 6278, Manises
  - Galderma Investigational Site 6295, Seville
  - Galderma Investigational Site 6311, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 53 study sites in 4 countries from 18 March 2022 to 04 January 2024.
Pre-assignment Details: A total of 258 participants were enrolled and treated in this study.
Groups:
- Nemolizumab 30 mg: Participants received a loading dose of 60 milligrams (mg) nemolizumab at Baseline followed by 2 subcutaneous (SC) injections for a total dose of 30 mg nemolizumab once every 4 weeks i.e. at Week 4 and Week 8.
- Nemolizumab 60 mg: Participants received 2 SC injections of 30 mg nemolizumab once every 4 weeks i.e. at Week 4 and Week 8.
Period: Overall Study
Arm/Group | Nemolizumab 30 mg | Nemolizumab 60 mg | Placebo
Started | 88 | 85 | 85
Completed | 72 | 71 | 72
Not Completed | 16 | 14 | 13
Not completed — Withdrawal by Subject | 5 | 3 | 4
Not completed — Adverse Event | 5 | 7 | 8
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Other-unspecified | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized participants.
Groups:
- Nemolizumab 30 mg: Participants received a loading dose of 60 mg nemolizumab at Baseline followed by 2 SC injections for a total dose of 30 mg nemolizumab once every 4 weeks i.e. at Week 4 and Week 8.
- Total: Total of all reporting groups
Arm/Group | Nemolizumab 30 mg | Nemolizumab 60 mg | Placebo | Total
Number analyzed (Participants) | 88 | 85 | 85 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (12.99) | 59.0 (13.00) | 58.4 (11.98) | 58.6 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 29 | 109
  Male | 47 | 46 | 56 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 31 | 40 | 113
  Not Hispanic or Latino | 46 | 54 | 45 | 145
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 3
  Asian | 3 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 21 | 32 | 24 | 77
  White | 56 | 43 | 50 | 149
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 6 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders With an Improvement of Worst Itch Numeric Rating Scale (WI NRS) Greater Than and Equal to (>=) 4 From Baseline at Week 12
Description: Responders are defined as participants with an improvement of >= 4 in WI NRS from baseline at Week 12 without use of rescue therapies and without treatment discontinuation due to lack of efficacy or Adverse event(AE)/death related to study drug. The WI NRS is a scale that is used by responders to report intensity of their worst pruritus (itch) during last 24 hours. Participants were asked following question: For worst itch intensity:"On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Higher scores indicated worse outcome. Percentage of responders with an improvement of WI NRS >= 4 from Baseline at Week 12 is reported here. Missing data due to discontinuation from the study prior to Week 12 or any other reason (e.g., insufficient eDiary completion) were imputed using multiple imputation under missing at random assumption (results were combined using Rubin's formulae).
Time Frame: Baseline, Week 12
Population: ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab 30 mg | Nemolizumab 60 mg | Placebo
Number analyzed (Participants) | 88 | 85 | 85
Percentage of Participants | 38.5 | 47.7 | 32.4
Statistical Analysis 1: Comparison: Nemolizumab 30 mg vs Placebo; Nemolizumab 30 mg versus Placebo; Test type: Superiority — Analysis was performed using hierarchical testing procedure. Testing was then performed sequentially in order the outcome measures were reported and continued when previous outcome measure was statistically significant at two-sided 0.025; p = 0.3696, Cochran-Mantel-Haenszel — Threshold of significance at 0.025; Strata adjusted percentage difference = 7.0, 97.5% CI 2-sided [-10.6 to 24.6]
Statistical Analysis 2: Comparison: Nemolizumab 60 mg vs Placebo; Nemolizumab 60 mg versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0686, Cochran-Mantel-Haenszel — Threshold of significance at 0.025; Strata adjusted percentage difference = 14.5, 97.5% CI 2-sided [-3.1 to 32.2]

2. Secondary Outcome: Percentage of Responders With an Improvement of WI NRS >= 3 From Baseline at Week 12
Description: Responders are defined as participants with an improvement of >= 3 in WI NRS from baseline at Week 12 without use of rescue therapies and without treatment discontinuation due to lack of efficacy or AE/death related to study drug. The WI NRS is a scale that is used by the responders to report the intensity of their worst pruritus (itch) during the last 24 hours. Participants were asked the following question: For worst itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Higher scores indicated worse outcome. Percentage of responders with an improvement of WI NRS >= 3 from Baseline at Week 12 is reported here. Missing data due to discontinuation from the study prior to Week 12 or any other reason (e.g., insufficient eDiary completion) were imputed using multiple imputation under missing at random assumption (results were combined using Rubin's formulae).
Time Frame: Baseline, Week 12
Population: ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab 30 mg | Nemolizumab 60 mg | Placebo
Number analyzed (Participants) | 88 | 85 | 85
Percentage of Participants | 49.3 | 60.6 | 47.1
Statistical Analysis 1: Comparison: Nemolizumab 30 mg vs Placebo; Analysis was performed using hierarchical testing procedure. Testing was then performed sequentially in order the outcome measures were reported and continued when previous outcome measure was statistically significant at two-sided 0.025; Test type: Superiority; p = 0.5909, Cochran-Mantel-Haenszel; Strata adjusted percentage difference = 4.3, 97.5% CI 2-sided [-13.8 to 22.3]
Statistical Analysis 2: Comparison: Nemolizumab 60 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1112, Cochran-Mantel-Haenszel; Strata adjusted percentage difference = 12.9, 97.5% CI 2-sided [-5.5 to 31.4]

3. Secondary Outcome: Percentage of Responders With an Improvement of WI NRS >= 4 From Baseline at Week 4
Description: Responders are defined as participants with an improvement of >= 4 in WI NRS from baseline at Week 4 without use of rescue therapies and without treatment discontinuation due to lack of efficacy or AE/death related to study drug. The WI NRS is a scale that is used by the responders to report the intensity of their worst pruritus (itch) during the last 24 hours. Participants were asked the following question: For worst itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Higher scores indicated worse outcome. Percentage of responders with an improvement of WI NRS >= 4 from Baseline at Week 4 is reported here. Missing data due to discontinuation from the study prior to Week 4 or any other reason (e.g., insufficient eDiary completion) were imputed using multiple imputation under missing at random assumption (results were combined using Rubin's formulae).
Time Frame: Baseline, Week 4
Population: ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab 30 mg | Nemolizumab 60 mg | Placebo
Number analyzed (Participants) | 88 | 85 | 85
Percentage of Participants | 24.3 | 26.6 | 7.4
Statistical Analysis 1: Comparison: Nemolizumab 30 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0034, Cochran-Mantel-Haenszel; Strata adjusted percentage difference = 17.3, 97.5% CI 2-sided [4.3 to 30.4]
Statistical Analysis 2: Comparison: Nemolizumab 60 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0025, Cochran-Mantel-Haenszel; Strata adjusted percentage difference = 17.1, 97.5% CI 2-sided [4.5 to 29.8]

4. Secondary Outcome: Percentage of Responders With an Improvement of Sleep Disturbance Numerical Rating Scale (SD NRS) >= 4 From Baseline at Week 12
Description: Responders are participants with an improvement >= 4 in SD NRS from baseline at Week 12 without use of rescue therapies and without treatment discontinuation due to lack of efficacy or AE/death related to study drug. SD NRS is a scale used by participants to report degree of their sleep loss related to chronic kidney disease with associated pruritus (CKD-aP ). Participants were asked following question: "On a scale of 0 to 10, with 0 being 'no sleep loss related to the symptoms of pruritus' and 10 being 'I did not sleep at all due to the symptoms of pruritus', how would you rate your sleep last night?". Higher scores indicated worse outcome. Percentage of responders with an improvement of SD NRS >= 4 from Baseline at Week 12 is reported here. Missing data due to discontinuation from study prior to Week 12 or any other reason (e.g., insufficient eDiary completion) were imputed using multiple imputation under missing at random assumption (results were combined using Rubin's formulae).
Time Frame: Baseline, Week 12
Population: ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab 30 mg | Nemolizumab 60 mg | Placebo
Number analyzed (Participants) | 88 | 85 | 85
Percentage of Participants | 27.7 | 42.6 | 25.3
Statistical Analysis 1: Comparison: Nemolizumab 30 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.5788, Cochran-Mantel-Haenszel; Strata adjusted percentage difference = 3.7, 97.5% CI 2-sided [-12.5 to 19.8]
Statistical Analysis 2: Comparison: Nemolizumab 60 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0303, Cochran-Mantel-Haenszel; Strata adjusted percentage difference = 16.5, 97.5% CI 2-sided [-0.8 to 33.9]

5. Secondary Outcome: Percentage of Responders With an Improvement of WI NRS >= 3 From Baseline at Week 4
Description: Responders are defined as participants with an improvement of >= 3 in WI NRS from baseline at Week 4 without use of rescue therapies and without treatment discontinuation due to lack of efficacy or AE/death related to study drug. The WI NRS is a scale that is used by the responders to report the intensity of their worst pruritus (itch) during the last 24 hours. Participants were asked the following question: For worst itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Higher scores indicated worse outcome. Percentage of responders with an improvement of WI NRS >= 3 from Baseline at Week 4 is reported here. Missing data due to discontinuation from the study prior to Week 4 or any other reason (e.g., insufficient eDiary completion) were imputed using multiple imputation under missing at random assumption (results were combined using Rubin's formulae).
Time Frame: Baseline, Week 4
Population: ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab 30 mg | Nemolizumab 60 mg | Placebo
Number analyzed (Participants) | 88 | 85 | 85
Percentage of Participants | 36.5 | 35.0 | 12.8
Statistical Analysis 1: Comparison: Nemolizumab 30 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel; Strata adjusted percentage difference = 24.2, 97.5% CI 2-sided [8.8 to 39.6]
Statistical Analysis 2: Comparison: Nemolizumab 60 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0021, Cochran-Mantel-Haenszel; Strata adjusted percentage difference = 20.8, 97.5% CI 2-sided [6.0 to 35.7]

6. Secondary Outcome: Percentage of Responders With an Improvement of SD NRS >= 4 From Baseline at Week 4
Description: Responders are defined as participants with an improvement >= 4 in SD NRS from baseline at Week 4 without use of rescue therapies and without treatment discontinuation due to lack of efficacy or AE/death related to study drug. The SD NRS is a scale used by participants to report the degree of their sleep loss related to CKD-aP. Participants were asked the following question: "On a scale of 0 to 10, with 0 being 'no sleep loss related to the symptoms of pruritus' and 10 being 'I did not sleep at all due to the symptoms of pruritus', how would you rate your sleep last night?". Higher scores indicated worse outcome. Percentage of responders with an improvement of SD NRS >= 4 from Baseline at Week 4 is reported here. Missing data due to discontinuation from the study prior to Week 4 or any other reason (e.g., insufficient eDiary completion) were imputed using multiple imputation under missing at random assumption (results were combined using Rubin's formulae).
Time Frame: Baseline, Week 4
Population: ITT population consisted of all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nemolizumab 30 mg | Nemolizumab 60 mg | Placebo
Number analyzed (Participants) | 88 | 85 | 85
Percentage of Participants | 16.1 | 23.6 | 2.8
Statistical Analysis 1: Comparison: Nemolizumab 30 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0028, Cochran-Mantel-Haenszel; Strata adjusted percentage difference = 14.0, 97.5% CI 2-sided [3.8 to 24.1]
Statistical Analysis 2: Comparison: Nemolizumab 60 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Strata adjusted percentage difference = 19.0, 97.5% CI 2-sided [7.6 to 30.5]

ADVERSE EVENTS:
Time Frame: From baseline up to Week 20
Description: Safety population included all participants who received at least one dose of the study drug.
Arm/Group | Nemolizumab 30 mg | Nemolizumab 60 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 4/86 | 4/84 | 5/85
Serious Adverse Events (participants affected / at risk) | 33/86 | 22/84 | 27/85
Other Adverse Events (participants affected / at risk) | 29/86 | 25/84 | 19/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nemolizumab 30 mg (N=86) | Nemolizumab 60 mg (N=84) | Placebo (N=85)
Pneumonia (Infections and infestations) | 2 | 1 | 5
Cellulitis (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 2
Abscess limb (Infections and infestations) | 0 | 0 | 1
Arteriovenous graft site infection (Infections and infestations) | 0 | 1 | 0
Bacterial myositis (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1
Candida pneumonia (Infections and infestations) | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 1
Cellulitis orbital (Infections and infestations) | 0 | 0 | 1
Chest wall abscess (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Diabetic foot infection (Infections and infestations) | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 1
Gangrene (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis clostridial (Infections and infestations) | 0 | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis acute (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 4 | 1 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 2
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1
Coronary artery aneurysm (Cardiac disorders) | 1 | 0 | 0
Coronary artery dissection (Cardiac disorders) | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 2 | 1 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous fistula maturation failure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic intracranial haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 4 | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 1 | 1
Syncope (Nervous system disorders) | 2 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Renal transplant (Surgical and medical procedures) | 1 | 1 | 2
Vascular access placement (Surgical and medical procedures) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Hypertensive urgency (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 1 | 0
Kidney transplant rejection (Immune system disorders) | 0 | 1 | 0
Liver transplant rejection (Immune system disorders) | 1 | 0 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Clear cell papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Post cardiac arrest syndrome (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nemolizumab 30 mg (N=86) | Nemolizumab 60 mg (N=84) | Placebo (N=85)
COVID-19 (Infections and infestations) | 1 | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2
Pneumonia (Infections and infestations) | 2 | 1 | 1
Bronchitis (Infections and infestations) | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 4 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 4
Toothache (Gastrointestinal disorders) | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 2
Eosinophilia (Blood and lymphatic system disorders) | 1 | 2 | 0
Polycythaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 3
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 3 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Dialysis hypotension (Vascular disorders) | 0 | 3 | 1
Hypotension (Vascular disorders) | 2 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT05075408/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT05075408/SAP_001.pdf